CLINICAL TRIAL: NCT04022967
Title: Randomized, Non-inferiority Trial Comparing a Dual Maintenance Therapy Strategy With Dolutegravir + Lamivudine (DTG/3TC) or Atazanavir/Ritonavir + Lamivudine (ATV/r+3TC) Versus the Standard WHO First Line Triple Therapy Tenofovir + Lamivudine + Efavirenz (TDF+3TC+EFV) or Dolutegravir + Lamivudine + Tenofovir (DTG+3TC+TDF) in West and Central African HIV-1 Infected Patients
Brief Title: ANRS 12372 MODERATO Study
Acronym: MODERATO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Mylan Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12372 MODERATO
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-05

CONDITIONS: HIV-1-infection
Keywords: Africa; Antiretroviral Treatment; HIV-1; Adults; Dual maintenance therapy; Dolutegravir; Atazanavir
MeSH Terms: interventions — dolutegravir; Ritonavir; Tenofovir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 : Dual maintenance therapy DTG+3TC (Experimental)
  Interventions: Drug: dolutegravir; Drug: Lamivudine
- Arm 2 : Dual maintenance therapy ATV/r+3TC (Experimental)
  Interventions: Drug: atazanavir boosted with ritonavir; Drug: Lamivudine
- Arm 3 : Reference triple therapy TDF+3TC+EFV or DTG+3TC+TDF (Active Comparator)
  Interventions: Drug: tenofovir + lamivudine +efavirenz or dolutegravir + lamivudine + tenofovir

INTERVENTIONS:
Drug: dolutegravir — One daily tablet (50mg) during 96 weeks
  Arms: Arm 1 : Dual maintenance therapy DTG+3TC
Drug: atazanavir boosted with ritonavir — One daily tablet with atazanavir (300 mg) boosted with ritonavir (100 mg) during 96 weeks
  Arms: Arm 2 : Dual maintenance therapy ATV/r+3TC
Drug: tenofovir + lamivudine +efavirenz or dolutegravir + lamivudine + tenofovir — One daily tablet with tenofovir 245 mg + lamivudine (300 mg) + efavirenz (400 mg) during 96 weeks OR One daily tablet with dolutegravir 50 mg + lamivudine (300 mg) + tenofovir (300 mg) during 96 weeks
  Arms: Arm 3 : Reference triple therapy TDF+3TC+EFV or DTG+3TC+TDF
Drug: Lamivudine — One daily tablet (300mg) during 96 weeks
  Arms: Arm 1 : Dual maintenance therapy DTG+3TC; Arm 2 : Dual maintenance therapy ATV/r+3TC

SUMMARY:
MODERATO is a phase III, open-label, randomized, multicenter, non-inferiority trial conducted in West and Central Africa (Cameroon, Côte d'Ivoire, Burkina Faso).

HIV-1 infected adults receiving first line ART with TDF+XTC+EFV or DTG+XTC+TDF virologically suppressed will be recruited and followed during 100 weeks.

The objective is to assess the non-inferiority of a strategy consisting of switching to a dual maintenance therapy (DTG+3TC or ATV/r+3TC), comparing to WHO standard first line regimen (TDF+3TC+EFV or DTG+3TC+TDF), in terms of virological success at 96 weeks

DETAILED DESCRIPTION:
In HIV-1 infected adults receiving first line ART with TDF+XTC+EFV or DTG+XTC+TDF virologically suppressed (viral load < detection limit of the technique used) for at least two years: to assess the non-inferiority of a strategy consisting of switching to a dual maintenance therapy (DTG+ 3TC or ATV/r+3TC), comparing to WHO standard first line regimen (TDF+3TC+EFV or DTG+3TC+TDF), in terms of virological success at 96 weeks, in Cameroon, Côte d'Ivoire and Burkina Faso.

This is a trial including two strategies (dual maintenance therapy and triple reference therapy) and three ART regimens (DTG+3TC and ATV/r+3TC used in the maintenance strategy and TDF+3TC+EFV/ DTG+3TC+TDF used in the reference strategy).

The primary analysis will compare the two strategies. Secondary analyses will compare the three ART regimens two by two.

In order to make these secondary analyses possible, participants will be randomly assigned, at inclusion, to each of the three ART regimens (arm 1: DTG+3TC; arm 2: ATV/r+3TC; arm 3: TDF+3TC+EFV / DTG+3TC+TDF). The maintenance strategy will include arm 1 and 2. The reference strategy will include arm 3

Number of participants : 480 (160 in each ART regimen, ie 320 in the dual maintenance therapy strategy and 160 in the triple therapy reference strategy)

The primary endpoint is treatment success, as defined by using the FDA snapshot algorithm : patients who are still continuing the assigned strategy and whose last available plasma HIV-1 RNA in the the window analysis (90 to 102 weeks) is <50 copies/ml at the end of the window analysis (90 to 102 weeks)

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Age of legal majority
* CD4 > 200 cells/mm3 at pre-inclusion
* Start first-line ART with non-nucleotide reverse transcriptase inhibitors including TDF+XTC+EFV for at least two years without a past history of virological failure, OR
* Be on TDF+XTC+EFV for at least two years then DTG+XTC+TDF without a past history of virological failure, OR
* Be on DTG+XTC+TDF (1st line regimen) for at least two years without a past history of virological failure
* Absence of past history of virological failure (viral load above the threshold corresponding to the test used); two blips between 50 and 200 copies/ml are allowed.
* At least 2 consecutive HIV-1 RNA < 50 copies/ml within past 2 years, including HIV-1 RNA at pre-inclusion
* Women with pregnancy potential are required to use an effective contraceptive method throughout the study follow up.
* Signed informed consent

Exclusion Criteria:

* HIV-2 infection or HIV-1+2 infection
* CD4 nadir <100 cells/mm3
* Chronic Hepatitis B (HBs Ag positive in the pre-inclusion balance)
* Ongoing active Tuberculosis
* Ongoing severe opportunistic infection
* Ongoing chemotherapy or immunotherapy
* Grade > 2 hemoglobin, neutrophil or platelet disorder
* ALT≥ 3 times the upper limit of normal value
* Creatinine clearance < 50 ml/min (CKD-EPI)
* Allergy to a trial drugs or drug component
* Ongoing pregnancy or Refusal of contraception
* Patient at risk of non-compliance
* Ongoing treatment with a drug that should not be associated with one of the drugs used in the study (cf appendix E page 77)
* Any symptoms or biological findings suggestive of a systemic disorder (renal, hepatic, cardiovascular, pulmonary) or other medical conditions that may interfere with the interpretation of test results or jeopardize the health of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2025-02-05 (Estimated); Study Completion 2025-02-05 (Estimated)

PRIMARY OUTCOMES:
The treatment success, as defined by using the FDA snapshot algorithm | 90 to 102 weeks
  Success : The proportion of patients who are still continuing the assigned strategy and whose last available plasma HIV-1 RNA in the the window analysis is <50 copies/ml at the end of the window analysis.
  Failure : patients who have discontinued the assigned strategy or whose last available plasma HIV-1 RNA in the window analysis (90 to 102 weeks) is ≥ 50 copies/ml or with no available HIV-1 RNA in the window analysis

SECONDARY OUTCOMES:
Failure combined endpoint | Between Day 0 and Week 96
  Percentage of participants who reach the following combined endpoint : "new drug-resistant resistance mutations observed", "decline of at least 20% in creatinine clearance" and "occurrence of at least one grade 3-4 neuropsychiatric disorder"
Plasma HIV-1 RNA | Between Day 0 and Week 96
  Evolution of plasma HIV-1 RNA
Virological success | Between Day 0 and Week 96
  Evolution of the percentage of participants with virological success (VL< 50 copies/Ml)
CD4 lymphocyte | Between Day 0 and Week 96
  Evolution of CD4 lymphocyte absolute count and percentage
Virological failure and new resistance mutations | Week 48 and Week 96
  Percentage of participants with virological failure and new resistance mutations
New HIV-1 drug resistance mutations | Week 48 and Week 96
  Profile of new HIV-1 drug resistance mutations observed in participants with virological failure
WHO stage 3-4 morbidity | Between Day 0 and Week 96
  Incidence of WHO stage 3-4 morbidity ( AIDS events and non AIDS severe morbidity)
ANRS grade 3-4 overall morbidity | Between Day 0 and Week 96
  Incidence of ANRS grade 3-4 overall morbidity (toxicity)
ANRS grade 3-4 renal morbidity | Between Day 0 and Week 96
  Incidence of ANRS grade 3-4 renal morbidity
ANRS grade 3-4 neurologic morbidity | Between Day 0 and Week 96
  Incidence of ANRS grade 3-4 neurologic morbidity
ANRS grade 3-4 hepatic morbidity | Between Day 0 and Week 96
  Incidence of ANRS grade 3-4 hepatic morbidity
Creatinine clearance | Between Day 0 and Week 96
  Evolution of creatinine clearance
Grade 1,2,3 or 4 renal disorders | Between Day 0 and Week 96
  Evolution of the percentage of patients with grade 1,2,3 or 4 renal disorders
Grade 1,2,3 or 4 hepatic liver disorders or abnormalities | Between Day 0 and Week 96
  Evolution of the percentage of patients with grade 1,2,3 or 4 hepatic liver disorders or abnormalities
Grade 1,2,3 or 4 CNS disorders | Between Day 0 and Week 96
  Evolution of the percentage of patients with grade 1,2,3 or 4 CNS disorders
Bone mineral density | Between Day 0 and Week 96
  Evolution of bone mineral density measured using CT bone density scan
Adherence to treatment using a self-questionnaire | Between Day 0 and Week 96
  Evolution of adherence to treatments measured using a self-questionnaire
Life quality | Between Day 0 and Week 96
  Evolution of quality of life measured using the ProQOL questionnaire
Symptoms | Between Day 0 and Week 96
  Evolution of symptoms using the "symptoms experienced" questionnaire
ARV drug plasma concentrations in participants with treatment failure | Between Day 0 and Week 96
  ARV drug plasma concentrations in participants with treatment failure
Switched back to triple therapy | Between Day 0 and Week 96
  Percentage of patients on dual therapy who switched back to triple therapy
Cost-effectiveness of the 3 ARV strategies | Week 96
  Cost-effectiveness of the 3 ARV strategies

CONTACTS AND LOCATIONS:
Overall Officials: Serge P. Eholié, MD, MSc, Pr, Principal Investigator — Service des Maladies Infectieuses et Tropicales, CHU de Treichville, Abidjan, Côte d'Ivoire; Roland Landman, MD, Principal Investigator — Institut de Médecine et d'Epidémiologie Appliquée - Hôpital Bichat Claude Bernard, Paris, France; Xavier Anglaret, MD, PhD, Study Director — Inserm 1219, Université de Bordeaux, France; Pierre-Marie Girard, MD, PhD, Study Chair — Infectious Diseases Department, University Hospital Saint Antoine, Paris, France
Locations (5):
- Burkina Faso (2):
  - Hôpital de jour, Service des maladies infectieuses, CHU Sourô Sanou, Bobo-Dioulasso
  - Service de médecine interne, CHU Yalgado Ouédraogo, Ouagadougou
- Service des Maladies Infectieuses, Hôpital du jour, Hôpital Central, Yaoundé, Cameroon
- Côte d’Ivoire (2):
  - Centre de Prise en Charge et de Formation (CePReF), Association ACONDA, Abidjan
  - Service des Maladies Infectieuses et Tropicales (SMIT), CHU de Treichville, Abidjan

REFERENCES:
- See also: Sponsor site — http://anrs.fr/
- See also: Related Info — http://www.mereva.net/